CLINICAL TRIAL: NCT05231369
Title: A Phase 1 Study to Evaluate Safety, Immunogenicity of the ChulaCov19 BNA159 mRNA Vaccine in Healthy Adults
Brief Title: Safety and Immunogenicity of ChulaCov19 BNA159 mRNA Vaccine
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chulalongkorn University (Other)
Collaborators: Chula Clinical Research Center (Chula CRC), Faculty of Medicine, Chulalongkorn University (Unknown); Academic Clinical Research Office (ACRO), Faculty of Medicine, Khon Kaen University (Unknown); BioNet-Asia (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: ChulaVac 003
Record Dates: First submitted 2022-02-07; First posted 2022-02-09 (Actual); Last update posted 2023-02-10 (Actual); Status verified 2023-02

CONDITIONS: Safety of 25 ug of ChulaCov19-BNA159 mRNA Vaccine; Tolerability of 25 ug of ChulaCov19-BNA159 mRNA Vaccine; Immune Response of 25 ug of ChulaCov19-BNA159 mRNA Vaccine; Safety of 50 ug of ChulaCov19-BNA159 mRNA Vaccine; Tolerability of 50 ug of ChulaCov19-BNA159 mRNA Vaccine; Immune Response of 50 ug of ChulaCov19-BNA159 mRNA Vaccine; Assess Which Dose is Appropriate to Use

STUDY DESIGN:
Intervention Model Description: If 25 ug dose is safe, then will proceed to enroll participants to receive 50 ug.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group 1: 25 ug of ChulaCov19 BNA159 mRNA vaccine (Experimental): The participants will receive 25 ug of the vaccine.
  Interventions: Biological: ChulaCov19 BNA159 mRNA vaccine
- group 2: 50 ug of ChulaCov19 BNA159 mRNA vaccine (Experimental): If 25 ug is safe, then will proceed to enroll 12 more participants to receive 50 ug.
  Interventions: Biological: ChulaCov19 BNA159 mRNA vaccine

INTERVENTIONS:
Biological: ChulaCov19 BNA159 mRNA vaccine — ChulaCov19 BNA159 mRNA vaccine is the lipid nanoparticles (LNPs)-encapsulated mRNA-based ChulaCov19 vaccine

SUMMARY:
This is a phase 1 study that will evaluate the safety and immunogenicity of ChulaCov19 BNA159 mRNA vaccine in healthy adults.

DETAILED DESCRIPTION:
ChulaCov19 BNA159 mRNA vaccine is the lipid nanoparticles (LNPs)-encapsulated mRNA-based ChulaCov19 vaccine developed by Chula VRC and manufactured by BioNet Asia, Thailand for the active immunisation of healthy adults against coronavirus disease 2019 (COVID-19). This is a phase 1 study that will evaluate the safety and immunogenicity of ChulaCov19 BNA159 mRNA vaccine in healthy adults. This study will be conducted in 2 study centers, open-label , dose finding, first in human (FIH) study conducted in healthy participants. There are two groups. One group will receive 25 ug of ChulaCov19 BNA159 mRNA vaccine and the other group will receive 50 ug of ChulaCov19 BNA159 mRNA vaccine. Each group will have 12 participants. Intramuscular injection of the investigational vaccine at the assigned dose, will be administered 21 days apart, on Day 1 and Day 22 ( ±3) .

ELIGIBILITY:
Inclusion Criteria:

1. Male or female participants between the ages of 18 and 60 years, inclusive, at enrolment
2. Women of child-bearing potential (WOCBP) may be enrolled in the study if the participant fulfils all the following criteria:

   1. Has a negative urine-based pregnancy test at screening and on the day of the first dose (Day1) and second dose (Day22)
   2. Must practice true abstinence or, if engaged in sexual relations with a male, they must agree to use highly effective (failure rate of < 1% per year when used consistently and correctly), double-barrier contraceptive measures* from screening and for a period of at least 60 days after the last dose of investigational vaccine.
   3. Is not currently breastfeeding.
3. Women of non-child-bearing potential may be enrolled in the study if the participant meet one of these following criteria:

   d. Postmenopausal (defined as having a history of amenorrhea of at least one year), or e. History of amenorrhea is less than one year, must have an FSH level > 40 milli-international units per milliliter (mIU/mL), or f. Have a documented status of being surgically sterile (hysterectomy, bilateral oophorectomy, or tubal ligation/salpingectomy).
4. Males must be surgically sterile (>30 days since vasectomy with no viable sperm), practice true abstinence or, if engaged in sexual relations with a female of child-bearing potential, the participants and their partner must use an acceptable, highly effective, double-barrier contraceptive method* from Screening and for a period of at least 60 days after the last dose of investigational vaccine.

   * The PI is to assess the adequacy of methods of contraception on a case-by-case basis. These criteria do not apply if the participants are in a same-sex relationship.

   Type of Participant and Disease Characteristics:
5. Participants must be able to communicate effectively with study personnel and agree to comply with the study procedures.
6. Capable to provide written informed consent.
7. Healthy participants who are determined by medical history, physical examination (if required), and clinical judgment of the investigator to be eligible for inclusion in the study.
8. Participants must have haematology, clinical chemistry, coagulation and urinalysis test results that are not deviating from the normal reference range by age and gender to a clinically relevant extent at Screening.

   Exclusion Criteria:
9. Presence of clinically significant medical history, unstable chronic or acute disease, or physical, or laboratory findings that, in the opinion of the PI may potentially increase the expected risk of exposure to the investigational vaccine, compromise the safety of the participant, or interfere with any aspect of study conduct or interpretation of results. This will include any thrombocytopenia or bleeding disorder contraindicating IM vaccination.
10. Known infection with human immunodeficiency virus (HIV), hepatitis C virus (HCV), or hepatitis B virus (HBV).
11. History of severe adverse reaction associated with a vaccine and/or severe allergic reaction (eg, anaphylaxis) to any component of the study intervention(s).
12. Participant has previously participated in an investigational study involving LNPs (a component of the investigational vaccine assessed in this trial).
13. Previous clinical (based on COVID-19 symptoms/signs alone, if a SARS-CoV-2 NAAT result was not available) or microbiological (based on COVID-19 symptoms/signs and a positive SARS-CoV-2 NAAT result) diagnosis of COVID-19.
14. Close contact with anyone known to have SARS-CoV-2 infection within 10 days prior to vaccine administration.
15. Individuals at high risk for severe COVID-19, including those with any of the following risk factors:

    * Uncontrolled hypertension
    * Diabetes mellitus
    * Cardiovascular disease
    * Chronic pulmonary disease
    * Asthma
    * Chronic liver disease
    * Stage 3 or worse chronic kidney disease (glomerular filtration rate <60 mL/min/1.73 m2)
    * BMI >30 kg/m2
    * Individuals with a history of autoimmune disease

    Prior/Concomitant Therapy:
16. Previous vaccination with any coronavirus vaccine at any time prior to the study or planned receipt of any other licensed or experimental SARS-CoV-2 vaccine within 50 days of receipt of the first study vaccination.
17. Receipt of medications intended to prevent COVID-19.
18. Chronic use (more than 14 continuous days) of or anticipated need to use, within the next 6 months, of any medications that may be associated with impaired immune responsiveness or with immunosuppression.
19. Receipt of immunoglobulins or blood products within 3 months of first vaccination.

    Diagnostic Assessments:
20. Positive on SAR-CoV-2 -RBD and/or -N antibody IgG/IgM at screening visit
21. Positive test for HIV, hepatitis B surface antigen (HBsAg) or hepatitis C virus antibodies (HCV Abs) at the screening visit.

    Other Exclusions:
22. Is a participant at high risk of SARS-CoV-2 exposure in the opinion of the PI (e.g., healthcare workers, active health care workers with direct patient contact, emergency response personnel).
23. Participation in other studies involving study intervention within 28 days prior to study entry and/or during study participation.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2022-12-14 (Actual); Primary Completion 2023-07-01 (Estimated); Study Completion 2023-07-01 (Estimated)

PRIMARY OUTCOMES:
Frequency of solicited local reactogenicity adverse events (AE) | during a 7-day follow-up period post each vaccination (up to Day 29+3)
  Frequency of solicited local reactogenicity adverse events (AE) during a 7-day follow-up period post each vaccination (up to Day 29+3)
Grade of solicited local reactogenicity adverse events (AE) | during a 7-day follow-up period post each vaccination (up to Day 29+3)
  Grade of solicited local reactogenicity adverse events (AE) during a 7-day follow-up period post each vaccination (up to Day 29+3)
Frequency of solicited systemic reactogenicity adverse events (AE) | during a 7-day follow-up period post each vaccination (up to Day 29+3)
  Frequency of solicited systemic reactogenicity adverse events (AE) during a 7-day follow-up period post each vaccination (up to Day 29+3)
Grade of solicited systemic reactogenicity adverse events (AE) | during a 7-day follow-up period post each vaccination (up to Day 29+3)
  Grade of solicited systemic reactogenicity adverse events (AE) during a 7-day follow-up period post each vaccination (up to Day 29+3)
Changes in vital signs | up to Visit 9 - Day 29 +3
  Changes in vital signs
Changes in physical examinations | up to Visit 9 - Day 29 +3
  Changes in physical examinations
Clinically relevant changes in laboratory measurement | up to Visit 9 - Day 29 +3
  Clinically relevant changes in laboratory measurement
Treatment-emergent, clinically significant changes in vital signs | up to Visit 9 - Day 29 +3
  Treatment-emergent, clinically significant changes in vital signs
Treatment-emergent, clinically significant changes in physical examinations | up to Visit 9 - Day 29 +3
  Treatment-emergent, clinically significant changes in physical examinations

SECONDARY OUTCOMES:
Frequency of unsolicited AEs | up to Day 50 ±3
  Frequency of unsolicited AEs
Grade of unsolicited AEs | up to Day 50 ±3
  Grade of unsolicited AEs
Frequency of SAEs | up to the end of the study Day387 ±14
  Frequency of SAEs
Frequency of MAAEs | up to the end of the study Day387 ±14
  Frequency of MAAEs
Frequency of NOCMCs | up to the end of the study Day387 ±14
  Frequency of NOCMCs
Geometric mean titres (GMT) | at Day29 (+3)
  SARS-Cov2-RBD-binding IgG antibody measured by enzyme-linked immunosorbent assay (ELISA)
Proportion of participants who achieved a greater than or equal to 4-fold rise from before vaccination to Day29 (+3) | before vaccination to Day29 (+3)
  SARS-Cov2-RBD-binding IgG antibody measured by enzyme-linked immunosorbent assay (ELISA)
Geometric mean ratio (GMR) defined as GMT ratio between the two doses of ChulaCov19 BNA159 mRNA vaccine | at Day29 (+3)
  SARS-Cov2-RBD-binding IgG antibody measured by enzyme-linked immunosorbent assay (ELISA)

OTHER OUTCOMES:
Geometric mean titres (GMT) | at Day 50 (±3)
  SARS-CoV-2- specific Pseudo-virus neutralization test with 50% inhibition titer (psVNT50) against wild type virus (WT)
Proportion of participants who achieved a greater than or equal to 4-fold rise from before vaccination to Day 50 (±3) | before vaccination to Day 50 (±3)
  SARS-CoV-2- specific Pseudo-virus neutralization test with 50% inhibition titer (psVNT50) against wild type virus (WT)
Geometric mean ratio (GMR) defined as GMT ratio between the two doses of ChulaCov19 BNA159 mRNA vaccine | at Day 50 (±3)
  SARS-CoV-2- specific Pseudo-virus neutralization test with 50% inhibition titer (psVNT50) against wild type virus (WT)
Geometric mean titres (GMT) | Day 29 (+3)
  SARS-CoV-2- specific Pseudo-virus neutralization test with 50% inhibition titer (psVNT50) against WT and variants of concern including Delta and Omicron
Geometric mean titres (GMT) | Day 50 (±3)
  SARS-CoV-2- specific Pseudo-virus neutralization test with 50% inhibition titer (psVNT50) against WT and variants of concern including Delta and Omicron
Geometric mean titres (GMT) | Day 112 (±7)
  SARS-CoV-2- specific Pseudo-virus neutralization test with 50% inhibition titer (psVNT50) against WT and variants of concern including Delta and Omicron
Geometric mean titres (GMT) | Day 202 (±7)
  SARS-CoV-2- specific Pseudo-virus neutralization test with 50% inhibition titer (psVNT50) against WT and variants of concern including Delta and Omicron
Geometric mean titres (GMT) | Day387 ±14
  SARS-CoV-2- specific Pseudo-virus neutralization test with 50% inhibition titer (psVNT50) against WT and variants of concern including Delta and Omicron
Proportion of participants who achieved a greater than or equal to 4-fold rise from before vaccination to Day 50 (±3) | before vaccination to Day 50 (±3)
  SARS-CoV-2- specific Pseudo-virus neutralization test with 50% inhibition titer (psVNT50) against WT and variants of concern including Delta and Omicron
Geometric mean ratio (GMR) defined as GMT ratio between the two doses of ChulaCov19 BNA159 mRNA vaccine | Day 29 (+3)
  SARS-CoV-2- specific Pseudo-virus neutralization test with 50% inhibition titer (psVNT50) against WT and variants of concern including Delta and Omicron
Geometric mean ratio (GMR) defined as GMT ratio between the two doses of ChulaCov19 BNA159 mRNA vaccine | Day 50 (±3)
  SARS-CoV-2- specific Pseudo-virus neutralization test with 50% inhibition titer (psVNT50) against WT and variants of concern including Delta and Omicron
Geometric mean ratio (GMR) defined as GMT ratio between the two doses of ChulaCov19 BNA159 mRNA vaccine | Day 112 (±7)
  SARS-CoV-2- specific Pseudo-virus neutralization test with 50% inhibition titer (psVNT50) against WT and variants of concern including Delta and Omicron
Geometric mean ratio (GMR) defined as GMT ratio between the two doses of ChulaCov19 BNA159 mRNA vaccine | Day 202 (±7)
  SARS-CoV-2- specific Pseudo-virus neutralization test with 50% inhibition titer (psVNT50) against WT and variants of concern including Delta and Omicron
Geometric mean ratio (GMR) defined as GMT ratio between the two doses of ChulaCov19 BNA159 mRNA vaccine | Day387 ±14
  SARS-CoV-2- specific Pseudo-virus neutralization test with 50% inhibition titer (psVNT50) against WT and variants of concern including Delta and Omicron
Geometric mean titres (GMT) | at Day 29 (+3)
  SARS-CoV-2- specific Live-virus neutralization test with 50% inhibition titer (MicroVNT50) against wild type virus (WT)
Geometric mean titres (GMT) | at Day 50 (±3)
  SARS-CoV-2- specific Live-virus neutralization test with 50% inhibition titer (MicroVNT50) against wild type virus (WT)
Proportion of participants who achieved a greater than or equal to 4-fold rise from before vaccination to Day 50 (±3) | before vaccination to Day 50 (±3)
  SARS-CoV-2- specific Live-virus neutralization test with 50% inhibition titer (MicroVNT50) against wild type virus (WT)
Geometric mean ratio (GMR) defined as GMT ratio between the two doses of ChulaCov19 BNA159 mRNA vaccine at Day 50 (±3) | at Day 50 (±3)
  SARS-CoV-2- specific Live-virus neutralization test with 50% inhibition titer (MicroVNT50) against wild type virus (WT)
Geometric mean titres (GMT) | at Day22
  SARS-CoV-2-surrogate viral neutralising antibody as measured by surrogate viral neutralising antibody assay (sVNT)
Geometric mean titres (GMT) | at Day 29 (+3)
  SARS-CoV-2-surrogate viral neutralising antibody as measured by surrogate viral neutralising antibody assay (sVNT)
Geometric mean titres (GMT) | at Day 50 (±3)
  SARS-CoV-2-surrogate viral neutralising antibody as measured by surrogate viral neutralising antibody assay (sVNT)
Geometric mean titres (GMT) | at Day 112 (±7)
  SARS-CoV-2-surrogate viral neutralising antibody as measured by surrogate viral neutralising antibody assay (sVNT)
Geometric mean titres (GMT) | at Day 202 (±7)
  SARS-CoV-2-surrogate viral neutralising antibody as measured by surrogate viral neutralising antibody assay (sVNT)
Geometric mean titres (GMT) | at Day387 ±14
  SARS-CoV-2-surrogate viral neutralising antibody as measured by surrogate viral neutralising antibody assay (sVNT)
Proportion of participants who achieved a greater than or equal to 4-fold rise from before vaccination to Day 50 (±3) | before vaccination to Day 50 (±3)
  SARS-CoV-2-surrogate viral neutralising antibody as measured by surrogate viral neutralising antibody assay (sVNT)
Geometric mean ratio (GMR) defined as GMT ratio between the two doses of ChulaCov19 BNA159 mRNA vaccine at Day 50 (±3) | at Day 50 (±3)
  SARS-CoV-2-surrogate viral neutralising antibody as measured by surrogate viral neutralising antibody assay (sVNT)
Geometric mean titres (GMT) | at Day22
  SARS-Cov2-RBD-binding IgG antibody measured by enzyme-linked immunosorbent assay (ELISA)
Geometric mean titres (GMT) | at Day 50 (±3)
  SARS-Cov2-RBD-binding IgG antibody measured by enzyme-linked immunosorbent assay (ELISA)
Geometric mean titres (GMT) | at Day 112 (±7)
  SARS-Cov2-RBD-binding IgG antibody measured by enzyme-linked immunosorbent assay (ELISA)
Geometric mean titres (GMT) | at Day 202 (±7)
  SARS-Cov2-RBD-binding IgG antibody measured by enzyme-linked immunosorbent assay (ELISA)
Geometric mean titres (GMT) | Day387 ±14
  SARS-Cov2-RBD-binding IgG antibody measured by enzyme-linked immunosorbent assay (ELISA)
Proportion of participants who achieved a greater than or equal to 4-fold rise from before vaccination to Day 50 (±3) | before vaccination to Day 50 (±3)
  SARS-Cov2-RBD-binding IgG antibody measured by enzyme-linked immunosorbent assay (ELISA)
Geometric mean ratio (GMR) defined as GMT ratio between the two doses of ChulaCov19 BNA159 mRNA vaccine at Day 50 (±3) | at Day 50 (±3)
  SARS-Cov2-RBD-binding IgG antibody measured by enzyme-linked immunosorbent assay (ELISA)
Geometric mean titres (GMT) of IgG | at Day22
  SARS-Cov2-spike protein-binding IgG antibody measured by enzyme-linked immunosorbent assay (ELISA)
Geometric mean titres (GMT) of IgG | at Day 29 (+3)
  SARS-Cov2-spike protein-binding IgG antibody measured by enzyme-linked immunosorbent assay (ELISA)
Geometric mean titres (GMT) of IgG | at Day 50 (±3)
  SARS-Cov2-spike protein-binding IgG antibody measured by enzyme-linked immunosorbent assay (ELISA)
Proportion of participants who achieved a greater than or equal to 4-fold rise from before vaccination to Day 50 (±3) | before vaccination to Day 50 (±3)
  SARS-Cov2-spike protein-binding IgG antibody measured by enzyme-linked immunosorbent assay (ELISA)
Geometric mean ratio (GMR) defined as GMT ratio between the two doses of ChulaCov19 BNA159 mRNA vaccine at Day 50 (±3) | at Day 50 (±3)
  SARS-Cov2-spike protein-binding IgG antibody measured by enzyme-linked immunosorbent assay (ELISA)
Percentage of participants who have positive specific T-cell IFNγ ELISpot responses (detectable above the assays cut-off) | on Day 29 (+3)
  SARS-CoV-2 spike protein-specific T-cell reposes as measured by IFNγ ELISpot assay
Percentage of participants who have positive specific T-cell IFNγ ELISpot responses (detectable above the assays cut-off) | on Day 50 (±3)
  SARS-CoV-2 spike protein-specific T-cell reposes as measured by IFNγ ELISpot assay
Percentage of participants who have positive specific T-cell IFNγ ELISpot responses (detectable above the assays cut-off) | on Day 112 (±7)
  SARS-CoV-2 spike protein-specific T-cell reposes as measured by IFNγ ELISpot assay
Percentage of participants who have positive specific T-cell IFNγ ELISpot responses (detectable above the assays cut-off) | on Day 202 (±7)
  SARS-CoV-2 spike protein-specific T-cell reposes as measured by IFNγ ELISpot assay
Median number of spot-forming cells (SFC) per 1 million PBMCs | on Day 29 (+3)
  SARS-CoV-2 spike protein-specific T-cell reposes as measured by IFNγ ELISpot assay
Median number of spot-forming cells (SFC) per 1 million PBMCs | on Day 50 (±3)
  SARS-CoV-2 spike protein-specific T-cell reposes as measured by IFNγ ELISpot assay
Median number of spot-forming cells (SFC) per 1 million PBMCs | on Day 112 (±7)
  SARS-CoV-2 spike protein-specific T-cell reposes as measured by IFNγ ELISpot assay
Median number of spot-forming cells (SFC) per 1 million PBMCs | on Day 202 (±7)
  SARS-CoV-2 spike protein-specific T-cell reposes as measured by IFNγ ELISpot assay
geometric mean of spot-forming cells (SFC) per 1 million PBMCs | on Day 29 (+3)
  SARS-CoV-2 spike protein-specific T-cell reposes as measured by IFNγ ELISpot assay
geometric mean of spot-forming cells (SFC) per 1 million PBMCs | on Day 50 (±3)
  SARS-CoV-2 spike protein-specific T-cell reposes as measured by IFNγ ELISpot assay
geometric mean of spot-forming cells (SFC) per 1 million PBMCs | on Day 112 (±7)
  SARS-CoV-2 spike protein-specific T-cell reposes as measured by IFNγ ELISpot assay
geometric mean of spot-forming cells (SFC) per 1 million PBMCs | on Day 202 (±7)
  SARS-CoV-2 spike protein-specific T-cell reposes as measured by IFNγ ELISpot assay
Percentage of participants who shows positive specific Th1 responses | on Day 29 (+3)
  SARS-CoV-2 spike protein-specific Th1/Th2 polarisation responses quantified by intracellular cytokine staining
Percentage of participants who shows positive specific Th1 responses | on Day 50 (±3)
  SARS-CoV-2 spike protein-specific Th1/Th2 polarisation responses quantified by intracellular cytokine staining
Median percentage specific Th1 responses, or Th2 response of each cohort | on Day 29 (+3)
  SARS-CoV-2 spike protein-specific Th1/Th2 polarisation responses quantified by intracellular cytokine staining
Median percentage specific Th1 responses, or Th2 response of each cohort | on Day 50 (±3)
  SARS-CoV-2 spike protein-specific Th1/Th2 polarisation responses quantified by intracellular cytokine staining

CONTACTS AND LOCATIONS:
Overall Officials: Sivaporn Gatechompol, MD, Principal Investigator — HIV-NAT, Thai Red Cross - AIDS Research Centre
Locations (2):
- Thailand (2):
  - Chula Clinical Research Center (Chula CRC), Faculty of Medicine, Chulalongkorn University, Bangkok
  - Academic Clinical Research Office (ACRO) Faculty of Medicine, Khon Kaen University, Khon Kaen